CLINICAL TRIAL: NCT06678971
Title: Effects of the 9-Week Warm-up Program, Basket Up, on Sports Performance in Young Basketball Athletes: A Randomized Controlled Trial
Brief Title: Effects of a Basketball-Specific Warm-Up, "Basket Up," on the Sports Performance of Young Basketball Players
Acronym: BASKETUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Collaborators: University of Valencia (Other)
Responsible Party: Principal Investigator, Juan F. Lisón Párraga, Dr, Professor, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNIVERSITY CARDENAL HERRERA-87
Record Dates: First submitted 2024-11-06; First posted 2024-11-07 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Jumping Performance; Speed; Agility
Keywords: Sports Performance; Speed; Agility; Jumping Performance; FIFA 11+; Warm-up; Basketball

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FIFA 11+ (Active Comparator): The intervention program takes place at the Alqueria del Basket facilities in Valencia, Spain, during the regular season. The warm-up regimen is supervised by a performance coach with expertise in basketball. Two days before the start of the program, athletes participate in an information and familiarization session. This session includes a verbal overview and a practical demonstration of the exercises, with the coach providing guidance and corrections to ensure athletes are well-prepared and able to perform the exercises correctly.
  The FIFA 11+ protocol consists of fifteen exercises organized into three segments, with three levels of difficulty. The first segment includes six running exercises, the second focuses on six exercises to enhance lower body strength, balance, and agility, and the third segment involves three running exercises aimed at activating the cardiovascular system.
  Interventions: Other: FIFA 11+
- Basket-Up (Experimental): The intervention program takes place at the Alqueria del Basket facilities in Valencia, Spain, during the regular season. The warm-up regimen is supervised by a performance coach with expertise in basketball. Two days before the start of the program, athletes participate in an information and familiarization session. This session includes a verbal overview and a practical demonstration of the exercises, with the coach providing guidance and corrections to ensure athletes are well-prepared and able to perform the exercises correctly.
  The Basket-Up warm-up program is developed by a committee of experts, including the medical staff and the Performance Department of Valencia Basket Club, with detailed information previously published. This protocol is specifically designed to address the physiological, functional, and physical demands of basketball training. It is structured into three phases with progressively increasing levels of difficulty, lasting a total of 20 minutes.
  Interventions: Other: Basket-Up

INTERVENTIONS:
Other: FIFA 11+ — The FIFA 11+ protocol consists of fifteen exercises organized into three segments, with three levels of difficulty. The first segment includes six running exercises, the second focuses on six exercises to enhance lower body strength, balance, and agility, and the third segment involves three running exercises aimed at activating the cardiovascular system.
  Arms: FIFA 11+
Other: Basket-Up — The Basket-Up warm-up program is developed by a committee of experts, including the medical staff and the Performance Department of Valencia Basket Club, with detailed information previously published. This protocol is specifically designed to address the physiological, functional, and physical demands of basketball training. Like the FIFA 11+ program, it is structured into three phases with progressively increasing levels of difficulty, lasting a total of 20 minutes.
  Phase 1 includes three exercises aimed at improving mobility. Phase 2 features six exercises focused on strength, direction changes, and plyometric activities. Phase 3 consists of six exercises designed to enhance agility and neurocognitive skills.
  Arms: Basket-Up

SUMMARY:
This study evaluates the effects of a specific 9-week basketball warm-up program, "BasketUp," on athletic performance, comparing it to the FIFA 11+ program. Male and female basketball players are randomly assigned to either the BasketUp or FIFA 11+ warm-up groups, performing these routines before practice three times a week for 9 weeks. Key performance metrics-sprinting speed, countermovement jump (CMJ), and agility-are measured at the start and end of the study.

DETAILED DESCRIPTION:
Current evidence is limited on the effectiveness of basketball-specific warm-up programs. This study evaluates the impact of a 9-week basketball-specific warm-up, "BasketUp," on sports performance, comparing it with the FIFA 11+ program. Male and female basketball athletes, are randomly assigned to either the BasketUp program or FIFA 11+. Both warm-ups are performed three times per week before basketball practice over the 9-week period. Performance measures-including sprinting, countermovement jump (CMJ), and agility-are assessed at the beginning and end of the intervention. A two-way mixed ANOVA analyzes the effect of time (baseline vs. 9 weeks) and group on these outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Have competed in at least one national basketball event within the past two years
* Consistently attend basketball practices throughout the season

Exclusion Criteria:

* Any current injury or condition restricting athletic activity
* A history of injury necessitating non-surgical treatment within the past 3 months
* A history of injury requiring surgery within the last 9 months

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Agility | At baseline and after 9 weeks
  We apply the Lane Agility Test (LAT), which is recognized as a basketball-specific test and is included in the National Basketball Association (NBA) Draft Combine tests. Its reliability is reported with a Cronbach's alpha coefficient of 0.973 and a coefficient of variation of 7.3%.
  For the test setup, four cones are placed at the corners of a designated area on the basketball court, forming a square. Participants complete the circuit as quickly as possible, incorporating sprints, lateral movements, and backward running. The time taken to complete the circuit is recorded with a handheld stopwatch. Each participant has two attempts, with a one-minute rest interval between them, and the best attempt is selected.
Vertical jump-related outcomes | At baseline and after 9 weeks
  The Countermovement Jump (CMJ) is chosen to analyze variables related to vertical jump performance. The portable ForceDecks pressure platform (ForceDecks, FDLite V.2, VALD, Brisbane, Australia) serves as the measurement instrument. The CMJ is one of the most commonly used evaluation methods for assessing lower-body explosive power, with strong reported reliability (Cronbach's alpha of 0.98 and a coefficient of variation of 2.4%).
  In this test, athletes start by standing on the platform with their hands on their waist. They are instructed to perform a maximum vertical jump by quickly transitioning from bent knees and hips to a fully extended position. Each participant has three attempts, with a 30-second rest interval between jumps, and the best attempt is selected. Data collected from this test include jump height and neuromuscular characteristics such as concentric and eccentric action times, asymmetrical distribution between legs, and jump power.
Velocity | At baseline and after 9 weeks
  We apply a 20-meter Sprint Test in which the athlete runs 20 meters at maximum speed. This test has demonstrated strong test-retest reliability, with a coefficient of 0.92.
  Athletes start in a standing position with their dominant foot forward. At the 20-meter mark, three photocells (Microgate® Polifemo Radio Light, Bolzano, Italy) are placed to record the athlete's time as they pass. Each participant has two attempts, with a one-minute rest interval between them, and the best attempt is selected.

CONTACTS AND LOCATIONS:
Locations (1):
- UCH CEU Univesity, Alfara del Patriarca, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided